CLINICAL TRIAL: NCT03379571
Title: Competing Risk of Death and End-stage Renal Disease in Incident Chronic Kidney Disease (Stages 3 to 5): the EPIRAN Community-based Study
Brief Title: Competing Risk of Death and ESRD in Incident CKD Patients
Acronym: EPIRAN
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: EPIRAN1
Record Dates: First submitted 2017-12-04; First posted 2017-12-20 (Actual); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Chronic Kidney Diseases
Keywords: Chronic kidney disease; Competing-risk analysis; Epidemiological study; Incidence; Outcomes; Risk factors
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Although chronic kidney disease (CKD) affects a growing number of people, epidemiologic data on incident CKD in the general population are scarce. Screening strategies to increase early CKD detection have been developed.

Methods: From a community-based sample of 4,409 individuals residing in a well-defined geographical area, investigators determined the number of patients having a first serum creatinine value ≥1.7 mg/dL and present for at least 3 months that allowed us to calculate an annual incidence rate of CKD (stages 3 to 5). CKD (stages 3 to 5) was defined by estimated glomerular filtration rate (eGFR) <60 mL/min/1.73 m2. Investigators also described the primary care, outcomes and risk factors associated with outcomes using competing risks analyses for these CKD patients.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years
* first serum creatinine value ≥1.7 mg/dL reached after January 1st, 2004
* and present for at least 3 months
* residing in the given geographical area (the Urban Community of Greater Nancy (UCGN))

Exclusion Criteria:

* <18 years
* prevalent CKD patient : CKD diagnosis before January 1st, 2004
* patients on dialysis or renal transplanted
* refusal of participation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population was incident CKD patients (stages 3 to 5) : all adult patients (≥18 years) residing in the given geographical area and having a first serum creatinine value ≥1.7 mg/dL reached after January 1st, 2004 and present for at least 3 months.
Sampling Method: Non-Probability Sample
Enrollment: 631 (Actual)
Dates: Start 2004-01-01 (Actual); Primary Completion 2009-12-31 (Actual); Study Completion 2009-12-31 (Actual)

PRIMARY OUTCOMES:
annual incidence rate of CKD | inclusion
  number of patients residing in a well-defined geographical area having a first serum creatinine value ≥1.7 mg/dL after January 1st, 2004 and still present for at least 3 months

SECONDARY OUTCOMES:
dialysis initiation | through study completion, 6 year after study start
  number of dialysis initiation.
death | through study completion, 6 year after study start
  number of death
management of CKD patients | through study completion, 6 year after study start
  %patients referred to a nephrologist, decline of the renal function

CONTACTS AND LOCATIONS:
Overall Officials: Michèle KESSLER, PU-PH, Principal Investigator — CHRU de Nancy

IPD SHARING:
Plan to Share IPD: No